CLINICAL TRIAL: NCT03721575
Title: Scarpa Fascia Preservation Versus Removal During Hernio-abdominoplasty: a Randomized Controlled Trial
Brief Title: Randomized Trial on Scarpa Fascia Preservation During Hernio-abdominoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura61
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scarpa's preserving hernio-abdominoplasty (Active Comparator): Hernio-abdominoplasty is performed with preservation of Scarpa's fascia.
  Interventions: Procedure: Scarpa's preserving hernio-abdominoplasty
- Classical hernio-abdominoplasty (Active Comparator): Hernio-abdominoplasty is performed with removalof Scarpa's fascia.
  Interventions: Procedure: Classical hernio-abdominoplasty

INTERVENTIONS:
Procedure: Scarpa's preserving hernio-abdominoplasty — Scarpa's fascia is preserved during hernio-abdominoplasty
  Arms: Scarpa's preserving hernio-abdominoplasty
Procedure: Classical hernio-abdominoplasty — Scarpa's fascia is removed during hernio-abdominoplasty
  Arms: Classical hernio-abdominoplasty

SUMMARY:
This randomized trial aimed to assess the efficacy of preservation of Scarpa's fascia during hernio-abdominoplasty in reducing the volume of postoperative drainage, accelerating time to drain removal and recovery, and reducing complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex ventral hernia that are fit for surgery (ASA class I and II) (Saklad, 1941).
* Patients with class III, IV according to Pitanguy's classification of abdominal deformities (Pitanguy, 1995).

Exclusion Criteria:

1. Patient with ASA class III, IV, and V.
2. Morbid obesity (BMI > 40).
3. Recurrent incisional hernias after mesh hernioplasty.
4. Strangulated hernias.
5. Isolated small paraumbilical hernias.
6. Patients with abdominal organomegaly and/or ascites.
7. Patients with coagulopathy,
8. Patients who are heavy smokers, patients with pulmonary problems, and patients with uncontrolled diabetes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Volume of postoperative drainage | Two weeks after surgery
  The volume of fluid drained through suction drains per 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, Principal Investigator — Mansoura University

IPD SHARING:
Plan to Share IPD: Undecided